CLINICAL TRIAL: NCT03961100
Title: A Randomized, Open-Label, Two Part Study to Explore the Performance of Entrectinib Prototype Mini-Tablet Formulations and the Effect of Drug Substance Particle Size On Entrectinib Bioavailability in Healthy Volunteers
Brief Title: A Performance and Bioavailability Study of Entrectinib in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP41341; 2019-000783-15 (EudraCT Number)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — entrectinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants will be randomly assigned to one of the three treatment sequences (T1T2R, T2RT1, RT1T2). In each treatment sequences, participants will cross-over to three periods taking different formulations of entrectinib. Entrectinib will be administered as a single 600 milligram (mg) oral dose under fed condition in three different formulations. Test formulation 1 (T1): film-coated mini-tablet; Test formulation 2 (T2): film-coated mini-tablet; Reference formulation (R): hard capsule.
  Interventions: Drug: Entrectinib 600 mg (T1); Drug: Entrectinib 600 mg (T2); Drug: Entrectinib 200 mg (R)
- Part 2 (Experimental): Participants will be randomly assigned to one of the two treatment sequences (TR, RT). In each treatment sequences, participants will cross-over to two periods taking different formulations of entrectinib. Entrectinib will be administered as a single 200 mg oral dose under fasted condition in two different formulations. Test formulation (T): hydroxypropyl methylcellulose (HPMC) capsule; Reference formulation (R): hard capsule.
  Interventions: Drug: Entrectinib 200 mg (R); Drug: Entrectinib 200 mg (T)

INTERVENTIONS:
Drug: Entrectinib 600 mg (T1) — Test formulation 1 (T1): Multi-particulate formulation 1: entrectinib film-coated mini-tablets
  Arms: Part 1
Drug: Entrectinib 600 mg (T2) — Test formulation 2 (T2): Multi-particulate formulation 2: entrectinib film-coated mini-tablets
  Arms: Part 1
Drug: Entrectinib 200 mg (R) — Reference formulation (R): entrectinib hard capsules
Drug: Entrectinib 200 mg (T) — Test formulation (T): entrectinib HPMC capsules
  Arms: Part 2

SUMMARY:
This study will evaluate the bioavailability, palatability, safety and tolerability of entrectinib in healthy volunteers. Part 1 of the study will explore the performance of entrectinib multi-particle formulation. Part 2 will evaluate the effect of drug substance particle size on entrectinib bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) between 18.0 and 32.0 kilogram per square meter (kg/m2), inclusive, and weighing >/=50 kg.
* Agreement to comply with measures to prevent pregnancy and restrictions on egg and sperm donation

Exclusion Criteria:

* Women of childbearing potential, women who are pregnant or breastfeeding, or intending to become pregnant during the study or within 14 days after the final dose of entrectinib or have a pregnant partner
* A clinical significant medical history of gastrointestinal surgery (e.g., gastric bypass) or other gastrointestinal disorder (e.g., malabsorption syndrome) that might affect absorption of medicines from the gastrointestinal tract
* Presence of a clinically significant disease, illness, medical condition or disorder, or any other medical history determined by the investigator to be clinically significant and relevant
* Clinically significant change in health status, or any major illness, or clinically significant acute infection or febrile illness
* Use of moderate or potent inhibitors or inducers of CYP P450 3A4 enzyme or P-gp transporter, or use of other prohibited medications
* Participation in any other clinical study involving an investigational medicinal product (IMP) or device
* A positive test result for hepatitis B, hepatitis C (HCV), or human immunodeficiency virus (HIV)
* Current smokers and those who have smoked, or users of e-cigarettes and nicotine replacement products within the last 12 months
* Known history of clinically significant hypersensitivity, or severe allergic reaction, to entrectinib or related compounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 T1T2R Sequence; Part 1 T2RT1 Sequence; Part 1 RT1T2 Sequence: Participants were randomly assigned to one of the three treatment sequences (T1T2R, T2RT1, RT1T2). In each treatment sequences, participants crossed over to three periods (each period=7 days) taking different formulations of entrectinib. Entrectinib was administered as a single 600 milligram (mg) oral dose under fed condition in three different formulations. Test formulation 1 (T1): film-coated mini-tablet; Test formulation 2 (T2): film-coated mini-tablet; Reference formulation (R): hard capsule. The washout period between entrectinib doses was at least 14 days.
- Part 2 TR Sequence; Part 2 RT Sequence: Participants were randomly assigned to one of the two treatment sequences (TR, RT). In each treatment sequences, participants crossed over to two periods (each period=7 days) taking different formulations of entrectinib. Entrectinib was administered as a single 200 mg oral dose under fasted condition in two different formulations. Test formulation (T): hydroxypropyl methylcellulose (HPMC) capsule; Reference formulation (R): hard capsule. The washout period between entrectinib doses was at least 14 days.
Period: Part 1
Arm/Group | Part 1 T1T2R Sequence | Part 1 T2RT1 Sequence | Part 1 RT1T2 Sequence | Part 2 TR Sequence | Part 2 RT Sequence
Started | 5 | 5 | 5 | 0 | 0
Completed | 5 | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 T1T2R Sequence | Part 1 T2RT1 Sequence | Part 1 RT1T2 Sequence | Part 2 TR Sequence | Part 2 RT Sequence
Started | 0 | 0 | 0 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 T1T2R Sequence | Part 1 T2RT1 Sequence | Part 1 RT1T2 Sequence | Part 2 TR Sequence | Part 2 RT Sequence | Total
Number analyzed (Participants) | 5 | 5 | 5 | 8 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (17.3) | 47.2 (15.2) | 39.8 (15.2) | 40.6 (11.5) | 46.8 (15.3) | 42.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 4 | 10
  Male | 4 | 3 | 4 | 6 | 4 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 5 | 5 | 4 | 6 | 8 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 5 | 5 | 8 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Entrectinib
Time Frame: At pre-defined intervals from study Day 1 to Day 5 of each periods (each period=7 days)
Population: The analysis population included all participants in Part 1 and Part 2, who received at least one dose of entrectinib. Only participants for whom data were collected are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Part 1 T1/F15 (Test Formulation 1); Part 1 T2/F16 (Test Formulation 2): Participants who received a single oral dose of 600 mg (240 × 2.5 mg) entrectinib film-coated mini-tablets in each period (one period=7 days) sprinkled on to, and mixed with, one tablespoon (15 mL) of yoghurt within 30 minutes of consumption of a standardized light "pediatric" breakfast. The washout period between entrectinib doses was at least 14 days.
- Part 1 R/F06 (Reference Formulation): Participants who received a single oral dose of 600 mg (3 × 200 mg) entrectinib hard capsule in each period (one period=7 days) swallowed whole with approximately 240 mL of water within 30 minutes of consumption of a standardized light "pediatric" breakfast. The washout period between entrectinib doses was at least 14 days.
- Part 2 T/F06 Coarse (Test Formulation): Participants who received a single oral dose of 1 x 200 mg entrectinib hydroxypropyl methylcellulose (HPMC) capsule in each period (one period=7 days) swallowed whole with approximately 240 mL of water after an overnight fast (minimum 8 hours). The washout period between entrectinib doses was at least 14 days.
- Part 2 R/F06 Fine (Reference Formulation): Participants who received a single oral dose of 1 x 200 mg entrectinib hard capsule in each period (one period=7 days) swallowed whole with approximately 240 mL of water after an overnight fast (minimum 8 hours). The washout period between entrectinib doses was at least 14 days.
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 16
nmol*h/L | 41500 (38.2) | 46600 (34.5) | 43400 (40.9) | 9860 (64.7) | 10100 (56.0)

2. Primary Outcome: AUC0-inf of Entrectinib Active Metabolite M5
Time Frame: At pre-defined intervals from study Day 1 to Day 5 of each periods (each period=7 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 16
nmol*h/L | 12400 (31.1) | 12200 (20.9) | 13600 (31.7) | 3900 (42.8) | 3780 (28.1)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Entrectinib
Time Frame: At pre-defined intervals from study Day 1 to Day 5 of each periods (each period=7 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 16
nmol/L | 1930 (24.9) | 1940 (21.3) | 1880 (26.1) | 494 (54.7) | 522 (33.8)

4. Primary Outcome: Cmax of Entrectinib Active Metabolite M5
Time Frame: At pre-defined intervals from study Day 1 to Day 5 of each periods (each period=7 days)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 16
nmol/L | 398 (32.2) | 325 (32.3) | 360 (30.1) | 100 (63.2) | 113 (42.4)

5. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Treatment-emergent adverse events (TEAEs) are AEs that were not present before the first dose of study drug or that were present before the first dose of study drug but worsened in intensity during exposure to study drug.
Time Frame: From Day -1 to Day 5 of each periods (each period=7 days)
Population: The analysis population included all participants in Part 1 and Part 2, who received at least one dose of entrectinib.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 16
Percentage of Participants | 100 | 93.3 | 100 | 31.3 | 37.5

ADVERSE EVENTS:
Time Frame: Day -1 through Day 5 of each period in both Part 1 and Part 2 (one period=7 days)
Description: The analysis population included all participants in Part 1 and Part 2, who received at least one dose of entrectinib.
Arm/Group | Part 1 T1/F15 (Test Formulation 1) | Part 1 T2/F16 (Test Formulation 2) | Part 1 R/F06 (Reference Formulation) | Part 2 T/F06 Coarse (Test Formulation) | Part 2 R/F06 Fine (Reference Formulation)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15 | 15/15 | 5/16 | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 T1/F15 (Test Formulation 1) (N=15) | Part 1 T2/F16 (Test Formulation 2) (N=15) | Part 1 R/F06 (Reference Formulation) (N=15) | Part 2 T/F06 Coarse (Test Formulation) (N=16) | Part 2 R/F06 Fine (Reference Formulation) (N=16)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 13 (13) | 11 (11) | 14 (14) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03961100/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03961100/SAP_001.pdf